CLINICAL TRIAL: NCT02515448
Title: A Pharmacokinetic-pharmacodynamic Dose Comparison Study of 8 mg/kg of Inhaled or Parenteral Gentamicin in 12 Mechanically Ventilated Critically Ill Patients Treated for Ventilator-associated Pneumonia
Acronym: GENTAERO
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GENTAERO
Record Dates: First submitted 2015-07-24; First posted 2015-08-04 (Estimated); Last update posted 2017-03-24 (Actual); Status verified 2016-05

CONDITIONS: Ventilator-associated Pneumonia
Keywords: VAP; Critical care; Pharmacokinetics; Gentamicin
MeSH Terms: conditions — Pneumonia, Ventilator-Associated | interventions — Gentamicins

ARMS (1):
- Gentamicine injectable(day 1+2)and then gentamicine inhalation (Experimental)
  Interventions: Drug: gentamicin

INTERVENTIONS:
Drug: gentamicin

SUMMARY:
Ventilator associated pneumonia (VAP) remains in the intensive care unit the infection associated with the highest morbidity and mortality.

Respiratory infection with resistant organism are increasing in prevalence. Because of lack of alternatives, amino glycoside, old antibiotics family, can be used for several infection.

Aerosolized Amikacin or Tobramycin are used in mechanically ventilated patients for respiratory infections. Gentamicin,which is effective against numerous multi drug resistant Gram-negative organism and Gram-positive like Staphylococcus aureus, could be a great option for nebulisation.

The investigators assume that nebulisation of gentamicin allows to obtain a higher lung concentration while assuring a systematic toxicity much lesser than a parenteral administration.

ELIGIBILITY:
Inclusion Criteria:

* to be in critical care unit
* to be mechanically ventilated
* to have a ventilator-associated pneumonia requiring a treatment by gentamicin
* to be affiliated to a national insurance scheme
* to have given an informed consent (patient or close person)

Exclusion Criteria:

* to be obese (BMI > 40 kg/m²)
* to have been treated by gentamicin for 7 days
* to be allergic to aminoglycoside
* to have a severe respiratory failure (PaO2 / FiO2 < 150)
* to have a renal failure (Cl creat < 60 ml/min/1.73m²)
* to be under reinforced protection measure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
"Peak Plasma Concentration (Cmax)" | 3 days

SECONDARY OUTCOMES:
PaO2/FiO2 ratio deterioration above 20%. | 3 days
  Bronchodilators used.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - BOISSON Matthieu, Poitiers, France
  - Dequin P-F, Tours, France